CLINICAL TRIAL: NCT02439398
Title: First-in-human, Double Blind, Randomized With Placebo, Open for the 6 First Patients (Dose Ranging) to Evaluate the Safety and Efficacy of Intracoronary Infusion of Allogeneic Human CSCs in Patients With AMI and Left Ventricular Dysfunction
Brief Title: Safety and Efficacy Evaluation of Intracoronary Infusion of Allogeneic Human Cardiac Stem Cells in Patients With AMI
Acronym: CAREMI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Coretherapix (Industry)
Collaborators: European Commission (Other); Universitaire Ziekenhuizen KU Leuven (Other); Saint-Louis Hospital, Paris, France (Other); Hospital General Universitario Gregorio Marañon (Other); Complejo Hospitalario de Navarra (Other); Hospital Clínico Universitario de Valladolid (Other); Hospital Donostia (Other); Hospital Clínico Universitario de Valencia (Other); University of Salamanca (Other); Hospital Universitario Virgen de la Victoria (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTPX01
Record Dates: First submitted 2015-04-27; First posted 2015-05-08 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Allogeneic human cardiac stem cells (Experimental): After randomization, subjects will received a suspension of allogeneic human cardiac stem cells (35 millions of CSCs - cell medicine) infused into the coronary artery responsible for the ischemic event.
  Interventions: Biological: Allogeneic human cardiac stem cells (CSCs)
- Placebo: Human Serum Albumin-HSA 5% (Placebo Comparator): After randomization, subjects will received placebo (which is also the cell medicine diluent). The placebo consists of a final administered volume of human serum albumin 5% in saline solution equivalent to the reconstituted cell medicine (18 mL). The placebo to be used is a marketed product (HSA 5%).
  Interventions: Other: Human Serum Albumin-HSA 5%

INTERVENTIONS:
Biological: Allogeneic human cardiac stem cells (CSCs) — Allogeneic human CSCs is a new cell medicine based on cells isolated from human heart biological samples (right atrium appendage of donors) and expanded in vitro.
  Other Names: AlloCSC-01
  Arms: Allogeneic human cardiac stem cells
Other: Human Serum Albumin-HSA 5% — Human Serum Albumin (HSA) is a well-known physiologic protein widely used in clinical practice and without known toxicity after parenteral administration.
  Arms: Placebo: Human Serum Albumin-HSA 5%

SUMMARY:
Development of myocardial reparative therapy for the treatment of acute ischemic cardiac disease, based on the intracoronary administration of allogeneic Cardiac Stem Cells (CSCs) to ameliorate myocardial cell death and promote cardio-regeneration.

The study comprises two phases:

1. Initial dose-escalation open-label safety phase comprising 6 patients. Escalation will start with the Maximum Recommended Safe Dose (MRSD) calculated from Non-Observed Adverse Events Level (NOAEL) and it is expected to finish with the target dose (TD). There will be no placebo group for this initial phase.
2. Randomized double-blind placebo-controlled safety and efficacy phase in which the TD will be injected if the dose-escalation phase is completed successfully.

DETAILED DESCRIPTION:
This is a "First in Patient" Clinical Trial to obtain safety and efficacy results about the intracoronary administration of a suspension of allogeneic cardiac stem cells (CSCs) for the treatment of ST elevation Myocardial Infarction (STEMI). This clinical trial will have a first dose-escalation phase in which the safety of 10, 20 and 35 million CSCs administration will be evaluated in 6 patients. A second double-blind randomized and placebo controlled phase will be initiated, if no major safety effects are observed during the first week after cell administration. The 35 million cells dose is the one expected to be used during the randomized phase.

Patients with EF<45% and with infarct sizes > 25% will be selected by magnetic resonance image (MRI). 49 patients will be included in the randomized phase with the aim of having 38 patients for efficacy analysis at the end of the follow up period (12 months). In this phase, patients will be randomly allocated for receiving CSCs or placebo in a 2:1 scheme. Three bioequivalent cellular batches obtained from different donors will be indistinctly used during the assay.

CSCs or placebo treatment will be infused into the coronary artery responsible for the ischemic event. Placebo will be a commercial preparation of human serum albumin 5% in saline solution that will also be used for cell product reconstitution.

After treatment, patients will be monitored overnight in a coronary care unit for any toxicity and discharged from hospital 24h after treatment if no adverse events are observed.

Subsequent safety follow-up will be done first at day 7 after treatment and then monthly or quarterly thereafter for 12 months. In addition, efficacy evaluations will be performed by MRI and clinical parameters at 1, 6 and 12 months after treatment.

Finally, cellular and humoral immunological response (screening for anti-HLA (Human Leukocyte Antigen) class I and class II antibodies, HLA typing, cross-matching between cells and treated patient and cytokine profiling in blood samples) will be analysed during the clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years of age and ≤ 80 years.
* Patients presenting a ST-segment-elevation myocardial infarction (STEMI) according to the universally accepted definition found in the STEMI management guide of the European Society of Cardiology
* Killip ≤ 2 on admission
* Successful primary coronary revascularization by Percutaneous Coronary Intervention- PCI - (Thrombolysis In Myocardial Infarction [TIMI] = 3) within 12h after the onset of infarct symptoms
* Bare-metal or drug-eluting stents (DES) of second generation (including new second generation stents, e.g. biolimus, novolimus and bioreabsorbable stents) at coronary revascularization by PCI
* Ejection Fraction (EF) ≤45% by magnetic resonance imaging (MRI). This MRI will be done between day 3 and day 5 after infarction and will be used as inclusion MRI
* Infarct size in left ventricle (LV) tested in the screening MRI ≥25% The presence of microvascular obstruction at inclusion MRI is permitted
* The affected coronary artery is adequate for cells infusion at the administration time. The administration procedure is technically feasible on day 4-7 after coronary revascularization by PCI
* The patient is stable and in adequate clinical condition to undergo the procedure.

Exclusion Criteria:

* Participation in another clinical trial in the last 30 days
* Previous allogeneic transplant (blood transfusions are allowed) or treated with cell or gene therapy
* Previous Q-wave infarction
* Significant valve disease, relapsing pericarditis, history of cardiac tamponade, cardiomyopathies
* Severe stenotic lesions (>90%) in a coronary vessel with size >2.75 mm not treated by PCI at least 24 hours before the baseline MRI study
* Previous EF≤45%, NYHA > 2 (New York Heart Association Functional Classification) or hospital admission for heart failure before STEMI
* Sustained VT that does not revert with treatment or requires >6 hours to be controlled in the 48 hours prior to the product administration procedure
* Complete atrioventricular blockade, or acute left bundle branch block in the 48 hours prior to the product administration procedure
* History of cardioembolic disease
* Platelets <100,000 and/or Hb<8.5g/dL
* Acute or chronic renal failure with creatinine ≥2.5 mg/dl or creatinine clearance ≤30 mL/min
* Infection with systemic involvement
* Cancer disease, except that eradicated at least 5 years before inclusion, and without receiving radiotherapy on chest. It is permitted coetaneous non-melanoma neoplasms completely eliminated (at any time) and that do not require subsequent chemotherapy or radiotherapy on chest.
* Child-Pugh's C stage chronic liver disease
* Baseline respiratory failure requiring oxygen at home
* Uncontrolled hypertension at screening despite treatment (systolic blood pressure [BP] ≥180 and/or diastolic BP ≥110)
* Very poorly controlled diabetes (Hb1Ac ≥8.5 g/dL) or with serious target organ lesion (peripheral vascular disease requiring revascularization or non revascularize)
* History of autoimmune disease
* Primary or acquired immune deficiency or immunosuppressant treatment (including treatments with immunosuppressants in the previous three months, or foreseeable need for those treatments during the course of the study).
* Women who are pregnant or breastfeeding or women of childbearing potential who do not agree to use contraceptives during the study period
* Life expectancy of less than 2 years for any reason.
* Allergy to aminoglycoside antibiotics or HSA hypersensitivity
* Contraindications preventing the use of Magnetic Resonance Imaging: Pacemaker, Implantable cardioverter-defibrillator (ICD), known reaction to gadolinium, claustrophobia, cochlear implants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Safety measured as the number of deaths and number of Major Adverse Cardiac Events (MACE) | 12 months
  The primary objective is to demonstrate the safety of the intra-coronary infusion of allogeneic cardiac stem cells in patients with a 7 days evolution first myocardial infarction and left ventricle dysfunction. Safety will be assessed a) evaluating the number of deaths from any cause within 30 days after cell medicine administration; b) evaluating the number of Major Adverse Cardiac Events (MACE) during the first 30 days (composite endpoint), defined as death from any cause, new Acute Myocardial Infarction (AMI), hospitalization due to Heart Failure (HF), sustained Ventricular Tachycardia (VT), Ventricular Fibrillation (VF), and stroke within 12 months after cell medicine administration.

SECONDARY OUTCOMES:
Efficacy measured by MRI as the infarct size change | 6 and 12 months
  Change of the Infarct Size as percentage (%) of LV mass analysed by MRI at 6 and 12 months after treatment administration versus screening MRI and 1 month MRI.
Efficacy measured by MRI as the evolution of biomechanical parameters | 6 and 12 months
  Percentage of change of the End Systolic Volume (ESV) and End Diastolic Volume (EDV), of the Wall Motion score as segmental contraction score, of the Sphericity Index, of the Systolic thickening by segment and of the Absolute change of Ejection Fraction (EF) analysed by MRI at 6 and 12 months after treatment administration versus screening MRI and 1 month MRI.
Efficacy measured by MRI as the evolution of edema | 1 month
  Percentage of change in the edema volume analysed by MRI at 1 month after treatment administration versus screening MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Paule Richard, MD, Study Director — Coretherapix (Tigenix Group)
Locations (1):
- Coretherapix (Tigenix Group), Tres Cantos, Madrid, Spain

REFERENCES:
- [Background] Boukouaci W, Lauden L, Siewiera J, Dam N, Hocine HR, Khaznadar Z, Tamouza R, Borlado LR, Charron D, Jabrane-Ferrat N, Al-Daccak R. Natural killer cell crosstalk with allogeneic human cardiac-derived stem/progenitor cells controls persistence. Cardiovasc Res. 2014 Nov 1;104(2):290-302. doi: 10.1093/cvr/cvu208. Epub 2014 Sep 11. PMID 25213554
- [Background] Lauden L, Boukouaci W, Borlado LR, Lopez IP, Sepulveda P, Tamouza R, Charron D, Al-Daccak R. Allogenicity of human cardiac stem/progenitor cells orchestrated by programmed death ligand 1. Circ Res. 2013 Feb 1;112(3):451-64. doi: 10.1161/CIRCRESAHA.112.276501. Epub 2012 Dec 12. PMID 23243206
- [Derived] Crisostomo V, Baez C, Abad JL, Sanchez B, Alvarez V, Rosado R, Gomez-Mauricio G, Gheysens O, Blanco-Blazquez V, Blazquez R, Toran JL, Casado JG, Aguilar S, Janssens S, Sanchez-Margallo FM, Rodriguez-Borlado L, Bernad A, Palacios I. Dose-dependent improvement of cardiac function in a swine model of acute myocardial infarction after intracoronary administration of allogeneic heart-derived cells. Stem Cell Res Ther. 2019 May 31;10(1):152. doi: 10.1186/s13287-019-1237-6. PMID 31151405
- [Derived] Fernandez-Aviles F, Sanz-Ruiz R, Bogaert J, Casado Plasencia A, Gilaberte I, Belmans A, Fernandez-Santos ME, Charron D, Mulet M, Yotti R, Palacios I, Luque M, Sadaba R, San Roman JA, Larman M, Sanchez PL, Sanchis J, Jimenez MF, Claus P, Al-Daccak R, Lombardo E, Abad JL, DelaRosa O, Corcostegui L, Bermejo J, Janssens S. Safety and Efficacy of Intracoronary Infusion of Allogeneic Human Cardiac Stem Cells in Patients With ST-Segment Elevation Myocardial Infarction and Left Ventricular Dysfunction. Circ Res. 2018 Aug 17;123(5):579-589. doi: 10.1161/CIRCRESAHA.118.312823. PMID 29921651
- [Derived] Sanz-Ruiz R, Casado Plasencia A, Borlado LR, Fernandez-Santos ME, Al-Daccak R, Claus P, Palacios I, Sadaba R, Charron D, Bogaert J, Mulet M, Yotti R, Gilaberte I, Bernad A, Bermejo J, Janssens S, Fernandez-Aviles F. Rationale and Design of a Clinical Trial to Evaluate the Safety and Efficacy of Intracoronary Infusion of Allogeneic Human Cardiac Stem Cells in Patients With Acute Myocardial Infarction and Left Ventricular Dysfunction: The Randomized Multicenter Double-Blind Controlled CAREMI Trial (Cardiac Stem Cells in Patients With Acute Myocardial Infarction). Circ Res. 2017 Jun 23;121(1):71-80. doi: 10.1161/CIRCRESAHA.117.310651. Epub 2017 May 22. PMID 28533209
- See also: Natural killer cell crosstalk with allogeneic human cardiac-derived stem/progenitor cells controls persistence. — http://www.ncbi.nlm.nih.gov/pubmed/25213554
- See also: Allogenicity of human cardiac stem/progenitor cells orchestrated by programmed death ligand — http://www.ncbi.nlm.nih.gov/pubmed/23243206
- See also: Sponsor web page — http://www.tigenix.com/
- See also: European Clinical Trial Data Base — https://www.clinicaltrialsregister.eu/ctr-search/search?query=Coretherapix